CLINICAL TRIAL: NCT05645211
Title: Agouti-related Peptide (AgRP) and the GH/IGF-1 Axis in Children
Brief Title: The AgRP and GH/IGF-1 Axis in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Pamela U. Freda, Professor of Medicine at CUIMC, Columbia University
Other Study IDs: AAAU4134
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Healthy children: 140 healthy children (70 females and 70 males) between the ages of 5-17 yr. will be studied; 7-8 children per year of this age range will be studied. They will be representative of the diverse racial and ethnic mix of children who receive their medical care at our medical center.
  Inclusion Criteria:
  1. Ambulatory male and female children aged 5-17 years
  2. Normal weight at birth
  3. Height between the 3rd and 99th percentiles of the mean as per the CDC growth percentiles.
  Exclusion Criteria:
  1. Genetic defects, chronic illnesses.
  2. Current prescription medication use
  3. Use of glucocorticoids, thyroid hormone or medications that may affect the GH-IGF-1 axis within 6 months of study entry.
- Group 2: Children with GH deficiency: 16 children (8 males, 8 females) between the ages of 5 - 9 yr. who are pre-pubertal and who plan to start GH treatment for isolated GH deficiency or idiopathic short stature.
  They will be representative of the diverse racial and ethnic mix of our hospital's patient population.
  GH deficiency:
  Inclusion Criteria:
  1. Ambulatory male and female children aged 5-9 years who are prepubertal
  2. Normal weight at birth
  3. Growth failure
  4. Peak GH response to 2 GH stimulation tests < 10 ng/ml
  5. Normal renal and liver function
  Exclusion criteria:
  1. Multiple pituitary hormone deficiencies,
  2. GH deficiency or poor growth associated with any acute or chronic medical condition such as renal disease or Turner's syndrome.
  3. History of diabetes or malignancy
  4. Use of glucocorticoids or medications known to affect the GH-IGF-1 axis within 6 months of study entry.
- Group 3: Children with short stature: Idiopathic Short Stature:
  Inclusion Criteria:
  1. Ambulatory male and female children aged 5-9 years who are prepubertal
  2. Normal weight at birth
  3. Height >2.25 SD below mean for age
  4. Peak GH response to 2 stimulation tests >10 ng/ml or normal IGF-1 and IGFBP-3 levels
  5. No prior supplemental growth hormone exposure
  6. Normal renal and liver function
  Exclusion criteria:
  1. Poor growth associated with any acute or chronic medical condition such as renal disease or Turner's syndrome.
  2. History of diabetes or malignancy
  3. Use of glucocorticoids or medications known to affect the GH-IGF-1 axis within 6 months of study entry.

SUMMARY:
Recent data support the existence of a GH-Agouti-related peptide (AgRP) axis. The neuropeptide AgRP promotes food intake and has important effects on energy homeostasis. Recent evidence suggest that GH stimulates AgRP and AgRP may mediate some of GH's important nutritional and metabolic effects. main goals of this project are to characterize, for the first time, plasma levels of AgRP in children and to determine how these relate to GH and IGF-1 levels, age, body composition, clinical and other endocrine parameters. To accomplish this, we will conduct two studies, one being a cross-sectional study that will measure AgRP levels in 140 healthy children ages 5-17 and the second being a prospective study that will measure the change in plasma AgRP levels in response to GH treatment in 16 children who receive this as part of their clinical care for GH deficiency or short stature.

DETAILED DESCRIPTION:
Protocol 1 This will be a cross-sectional study in 140 healthy children. Participation will include one visit that will take place between 8-9 am and after a fast from midnight the night before.

Procedures at the visit will include:

1. Review of medical history
2. Anthropometrics measurements: Weight, height, waist and hip circumferences.
3. Collection of information from medical record including growth records and physical examination findings including features relevant to pubertal stage in all children and onset of menses in females.
4. Assessment of pubertal status and Tanner stage based on physical examination.
5. Collection of information on diet, activity level and sleep.
6. Blood Sampling: venous blood will be sampled from a peripheral vein for measurement of AgRP, GH, IGF-1, leptin, SOb-R, triglycerides, insulin, glucose, testosterone(males), estradiol(females), DHEAS and cortisol levels. Insulin and glucose levels will be used to assess insulin resistance by HOMA & QUICKI.

Protocol 2 This will be a prospective study in 16 children who will be studied before and at 4 time points (1 week, 2 weeks, 1 month and 2 months) after starting GH treatment as part of their clinical care. This protocol will study subjects Groups 2 and 3. Growth hormone will not be prescribed as part of this study. Children will be treated clinically with GH as prescribed by their Pediatric Endocrinologist for FDA approved indications and according to standard guidelines for dosing for treatment of GH deficiency in children.

Each visit that will take place between 8-9 am and after a fast from midnight the night before.

Procedures at each visit will include:

1. Review of medical history
2. Anthropometrics measurements: Weight, height, waist and hip circumferences, skinfold thicknesses.
3. Collection of information from medical record including growth records and physical examination findings including features relevant to pubertal stage in all children and onset of menses in females. GH dose and compliance will be recorded at follow up visits.
4. Collection of information on diet, activity level and sleep.
5. Blood Sampling: Venous blood will be sampled at a peripheral vein for:

Baseline (pre-GH treatment): measurement of AgRP, GH, IGF-1, IGFBP-3, leptin, SOb-R, triglycerides, insulin and glucose, testosterone(males), estradiol(females), DHEAS and cortisol levels.

Follow up visits on growth hormone: measurement of AgRP, IGF-1, IGFBP-3, leptin, SOb-R, triglycerides, insulin, glucose and cortisol levels.

Insulin and glucose levels will be used to assess insulin resistance by HOMA & QUICKI.

ELIGIBILITY:
Healthy children

Inclusion Criteria:

1. Ambulatory male and female children aged 5-17 years
2. Normal weight at birth
3. Height between the 3rd and 99th percentiles of the mean as per the CDC growth percentiles.

Exclusion Criteria:

1. Genetic defects, chronic illnesses.
2. Current prescription medication use
3. Use of glucocorticoids, thyroid hormone or medications that may affect the GH-IGF-1 axis within 6 months of study entry.

Children with GH deficiency:

Inclusion Criteria:

1. Ambulatory male and female children aged 5-9 years who are prepubertal
2. Normal weight at birth
3. Growth failure
4. Peak GH response to 2 GH stimulation tests < 10 ng/ml
5. Normal renal and liver function

Exclusion criteria:

1. Multiple pituitary hormone deficiencies,
2. GH deficiency or poor growth associated with any acute or chronic medical condition such as renal disease or Turner's syndrome.
3. History of diabetes or malignancy
4. Use of glucocorticoids or medications known to affect the GH-IGF-1 axis within 6 months of study entry.

Children with idiopathic Short Stature:

Inclusion Criteria:

1. Ambulatory male and female children aged 5-9 years who are prepubertal
2. Normal weight at birth
3. Height >2.25 SD below mean for age
4. Peak GH response to 2 stimulation tests >10 ng/ml or normal IGF-1 and IGFBP-3 levels
5. No prior supplemental growth hormone exposure
6. Normal renal and liver function

Exclusion criteria:

1. Poor growth associated with any acute or chronic medical condition such as renal disease or Turner's syndrome.
2. History of diabetes or malignancy
3. Use of glucocorticoids or medications known to affect the GH-IGF-1 axis within 6 months of study entry.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children: 140 healthy children (70 females and 70 males) between the ages of 5-17 yr. will be studied; 7-8 children per year of this age range will be studied. They will be representative of the diverse racial and ethnic mix of children who receive their medical care at our medical center.Children will be recruited from among the healthy children visiting primary care Pediatricians at our medical center.
  GH deficient and idiopathic short stature children: 16 children (8 males, 8 females) between the ages of 5 - 9 yr. who are pre-pubertal and who plan to start GH treatment for isolated GH deficiency or idiopathic short stature. They will be representative of the diverse racial and ethnic mix of our hospital's patient population.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2026-06-10 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Protocol 1: Correlation of Plasma AgRP levels with IGF-1 levels | Baseline (cross-sectional at single time point, no intervention)
  Plasma AgRP levels correlation with IGF-1 levels Protocol 1: Correlation of Plasma AgRP levels with IGF-1 levels
Protocol 2: Change in plasma AgRP levels with GH therapy | baseline to 2 months
  Change in plasma AgRP levels from pre-GH therapy to post-GH therapy

SECONDARY OUTCOMES:
Protocol 1: Correlation of plasma AgRP levels with age | Baseline (cross-sectional testing at one time point, no intervention)
  Correlation of plasma AgRP levels with age
Protocol 1: Correlation of plasma AgRP levels with leptin levels | Baseline (cross-sectional testing at one time point, no intervention)
  Correlation of plasma AgRP levels with leptin levels
Protocol 1: Correlation of plasma AgRP with percent body fat (determined from skinfold thickness) | Baseline (cross-sectional testing at one time point, no intervention)
  Correlation of plasma AgRP with percent body fat (determined from skinfold thickness)
Protocol 2: Change in AgRP levels correlation with change in IGF-1 levels | Baseline to 2 months
  Correlation of change in AgRP levels with change in IGF-1 levels from baseline to 2 months of GH therapy
Protocol 2: Change in AgRP level correlation with pre-treatment leptin levels | Baseline to 2 months
  Correlation of change in AgRP level from baseline to 2 months of GH therapy with pre-treatment leptin levels

IPD SHARING:
Plan to Share IPD: No